CLINICAL TRIAL: NCT00388167
Title: PROCAS: Study Observational Prospective and Multicenter to Determine the Clinic Effectiveness and the Safety of Caspofungin Acetate (CANCIDAS®) in the Treatment of Invader Fungal Infection
Brief Title: Acetato de Caspofungin (Cancidas®) in the Treatment of Fungal Infection
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Collaborators: GTEI (Unknown); SEMICYUC (Unknown)
Responsible Party: Pethema, pethema
Other Study IDs: PET-CAS-2003-01; PET-CAS-2004-01
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Candidiasis; Aspergillosis
Keywords: Invader fungal infection (IFI); Invasive Aspergillosis (AI); Invasive Candidiasis (CI); Caspofungin acetate
MeSH Terms: conditions — Candidiasis; Aspergillosis; Candidiasis, Invasive | interventions — Caspofungin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Caspofungin
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — The patients are treated with 70 mg IV of caspofungin on day 1, followed by 50 mg/day IV during the rest of treatment

SUMMARY:
We wanted to determine the efficacy and the safety of caspofungin acetate (CANCIDAS®) in the treatment of invader fungal infection (IFI) specifically, Invasive Candidiasis (CI) in adults patients without neutropenia and Invasive Aspergillosis (AI) in adults patients who are refractory to or intolerant of other therapies (i.e., amphotericin B, lipid formulations of amphotericin B, and/or itraconazole).

DETAILED DESCRIPTION:
Study post-marketing (observational). It is multicenter and prospective. No masking is used, without control group neither is randomized

ELIGIBILITY:
Inclusion Criteria:

* Female and male with 18 years old at least.
* Diagnosis of AI or CI. It will be based in Clinical History, signs and symptoms that the patient takes, discovery of studies of radiology and results of cultivation and/or studies of anatomopathology positives for Candida spp. or Aspergillus spp.
* Patients with AI, must be refractory to or intolerant of other therapies antifungal used in the hospital.
* Patients with CI, must be or not refractory to or intolerant of other therapies antifungal used in the hospital.

Exclusion Criteria:

* Patients with diagnosis uncertain based in one or more of next criterions: Cultivation positive for Candida in an only localization (urine, spittle, end/current of catheter; osteomyelitis or endocarditis by Candida without treatment appropriated surgical; infection by Candida of prosthetic material without retired of the same; positive blood cultive for Candida in appearance of vascular prosthesis; allergic lung Aspergillosis; and aspergilloma or aspergillosis eye without treatment appropriated surgical).
* Allergic / hypersensitivity to caspofungin.
* Insufficiency several liver (rate of Chile-Pugh >9).
* Prediction of survival <5 days.
* Pregnant or breast feeding.
* Previous Participation of patient in this study.
* Presence of other disease or any condition that it can mix up the interpretation of results or create risks.
* Previous Participation of patient in other clinical study that it involve the administration of a drug in investigation in the 14 days previous to your inclusion in the study or during the administration of caspofungin. We can include patients took with antineoplastic drugs in research whenever at lefts a Investigator Coordinator authorizes it before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of AI or CI
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2004-03; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Sanz, Dr, Principal Investigator — Hospital La Fe
Locations (27):
- Spain (27):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital vall d'Hebrón, Barcelona, Barcelona
  - Institut Català d'Oncología, L'Hospitalet de Llobregat, Barcelona
  - Xarxa assistencial de Manresa, Manresa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Complejo Hospitalario Xeral-Cies, Vigo, Vigo
  - Area Hospitalaria Juan Ramón Jimenez, Huelva
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera

REFERENCES:
- [Background] Keating GM, Jarvis B. Caspofungin. Drugs. 2001;61(8):1121-9; discussion 1130-1. doi: 10.2165/00003495-200161080-00007. PMID 11465873
- [Background] Tkacz JS. Glucan biosynthesis in fungi and its inhibition. In: Sutcliff JA, Georgopapadaku NH, eds. Emerging Targets in Antibacterial and Antifungal Chemotherapy. New York: Routledge, Chapman & Hall, 1992; 495-523.
- [Background] Groll AH, Walsh TJ. Potential new antifungal agents. Curr Opin Infect Dis 1997; 10: 449-458
- [Background] Debono M, Gordee RS. Antibiotics that inhibit fungal cell wall development. Annu Rev Microbiol. 1994;48:471-97. doi: 10.1146/annurev.mi.48.100194.002351. PMID 7826015
- [Background] Denning DW. Echinocandins and pneumocandins--a new antifungal class with a novel mode of action. J Antimicrob Chemother. 1997 Nov;40(5):611-4. doi: 10.1093/jac/40.5.611. No abstract available. PMID 9421307
- [Background] Arikan S, Lozano-Chiu M, Paetznick V, Rex JH. In vitro synergy of caspofungin and amphotericin B against Aspergillus and Fusarium spp. Antimicrob Agents Chemother. 2002 Jan;46(1):245-7. doi: 10.1128/AAC.46.1.245-247.2002. PMID 11751145
- [Background] Graybill JR, Najvar LK, Luther MF, Fothergill AW. Treatment of murine disseminated candidiasis with L-743,872. Antimicrob Agents Chemother. 1997 Aug;41(8):1775-7. doi: 10.1128/AAC.41.8.1775. PMID 9257759
- [Background] Espinel-Ingroff A. Comparison of In vitro activities of the new triazole SCH56592 and the echinocandins MK-0991 (L-743,872) and LY303366 against opportunistic filamentous and dimorphic fungi and yeasts. J Clin Microbiol. 1998 Oct;36(10):2950-6. doi: 10.1128/JCM.36.10.2950-2956.1998. PMID 9738049
- [Background] Bartizal K, Gill CJ, Abruzzo GK, Flattery AM, Kong L, Scott PM, Smith JG, Leighton CE, Bouffard A, Dropinski JF, Balkovec J. In vitro preclinical evaluation studies with the echinocandin antifungal MK-0991 (L-743,872). Antimicrob Agents Chemother. 1997 Nov;41(11):2326-32. doi: 10.1128/AAC.41.11.2326. PMID 9371328
- [Background] Kurtz MB, Heath IB, Marrinan J, Dreikorn S, Onishi J, Douglas C. Morphological effects of lipopeptides against Aspergillus fumigatus correlate with activities against (1,3)-beta-D-glucan synthase. Antimicrob Agents Chemother. 1994 Jul;38(7):1480-9. doi: 10.1128/AAC.38.7.1480. PMID 7979276
- [Background] Arikan S, Lozano-Chiu M, Paetznick V, Rex JH. In vitro susceptibility testing methods for caspofungin against Aspergillus and Fusarium isolates. Antimicrob Agents Chemother. 2001 Jan;45(1):327-30. doi: 10.1128/AAC.45.1.327-330.2001. PMID 11120990
- [Background] Bowman JC, Hicks PS, Kurtz MB, Rosen H, Schmatz DM, Liberator PA, Douglas CM. The antifungal echinocandin caspofungin acetate kills growing cells of Aspergillus fumigatus in vitro. Antimicrob Agents Chemother. 2002 Sep;46(9):3001-12. doi: 10.1128/AAC.46.9.3001-3012.2002. PMID 12183260
- [Background] Pfaller MA, Marco F, Messer SA, Jones RN. In vitro activity of two echinocandin derivatives, LY303366 and MK-0991 (L-743,792), against clinical isolates of Aspergillus, Fusarium, Rhizopus, and other filamentous fungi. Diagn Microbiol Infect Dis. 1998 Apr;30(4):251-5. doi: 10.1016/s0732-8893(97)00246-0. PMID 9582584
- [Background] Del Poeta M, Schell WA, Perfect JR. In vitro antifungal activity of pneumocandin L-743,872 against a variety of clinically important molds. Antimicrob Agents Chemother. 1997 Aug;41(8):1835-6. doi: 10.1128/AAC.41.8.1835. PMID 9257774
- [Background] Scott Hicks P, Dorso K, Gerckens I, et al. Comparative In Vitro Susceptibility of Clinical Trial Isolates to the Echinocandin Antifungal Caspofungin (Cancidas, MK- 0991) (Abstract: 193). 40th Interscience Conference on Antimicrobial Agents and Chemotherapy, Toronto (Canada), 2000.
- [Background] Barchiesi F, Schimizzi AM, Fothergill AW, Scalise G, Rinaldi MG. In vitro activity of the new echinocandin antifungal, MK-0991, against common and uncommon clinical isolates of Candida species. Eur J Clin Microbiol Infect Dis. 1999 Apr;18(4):302-4. doi: 10.1007/pl00015011. PMID 10385023
- [Background] Marco F, Pfaller MA, Messer SA, Jones RN. Activity of MK-0991 (L-743,872), a new echinocandin, compared with those of LY303366 and four other antifungal agents tested against blood stream isolates of Candida spp. Diagn Microbiol Infect Dis. 1998 Sep;32(1):33-7. doi: 10.1016/s0732-8893(98)00050-9. PMID 9791755
- [Background] Vazquez JA, Lynch M, Boikov D, Sobel JD. In vitro activity of a new pneumocandin antifungal, L-743,872, against azole-susceptible and -resistant Candida species. Antimicrob Agents Chemother. 1997 Jul;41(7):1612-4. doi: 10.1128/AAC.41.7.1612. PMID 9210698
- [Background] Krishnarao TV, Galgiani JN. Comparison of the in vitro activities of the echinocandin LY303366, the pneumocandin MK-0991, and fluconazole against Candida species and Cryptococcus neoformans. Antimicrob Agents Chemother. 1997 Sep;41(9):1957-60. doi: 10.1128/AAC.41.9.1957. PMID 9303393
- [Background] Nelson PW, Lozano-Chiu M, Rex JH. In vitro growth-inhibitory activity of pneumocandins L-733,560 and L-743,872 against putatively amphotericin B- and fluconazole-resistant Candida isolates: influence of assay conditions. J Med Vet Mycol. 1997 Jul-Aug;35(4):285-7. PMID 9292427
- [Background] Pfaller MA, Messer SA, Gee S, Joly S, Pujol C, Sullivan DJ, Coleman DC, Soll DR. In vitro susceptibilities of Candida dubliniensis isolates tested against the new triazole and echinocandin antifungal agents. J Clin Microbiol. 1999 Mar;37(3):870-2. doi: 10.1128/JCM.37.3.870-872.1999. PMID 9986880
- [Background] Douglas CM, D'Ippolito JA, Shei GJ, Meinz M, Onishi J, Marrinan JA, Li W, Abruzzo GK, Flattery A, Bartizal K, Mitchell A, Kurtz MB. Identification of the FKS1 gene of Candida albicans as the essential target of 1,3-beta-D-glucan synthase inhibitors. Antimicrob Agents Chemother. 1997 Nov;41(11):2471-9. doi: 10.1128/AAC.41.11.2471. PMID 9371352
- [Background] Kurtz MB, Abruzzo G, Flattery A, Bartizal K, Marrinan JA, Li W, Milligan J, Nollstadt K, Douglas CM. Characterization of echinocandin-resistant mutants of Candida albicans: genetic, biochemical, and virulence studies. Infect Immun. 1996 Aug;64(8):3244-51. doi: 10.1128/iai.64.8.3244-3251.1996. PMID 8757860
- [Background] Douglas CM, Marrinan JA, Li W, Kurtz MB. A Saccharomyces cerevisiae mutant with echinocandin-resistant 1,3-beta-D-glucan synthase. J Bacteriol. 1994 Sep;176(18):5686-96. doi: 10.1128/jb.176.18.5686-5696.1994. PMID 8083161
- [Background] Osherov N, May GS, Albert ND, Kontoyiannis DP. Overexpression of Sbe2p, a Golgi protein, results in resistance to caspofungin in Saccharomyces cerevisiae. Antimicrob Agents Chemother. 2002 Aug;46(8):2462-9. doi: 10.1128/AAC.46.8.2462-2469.2002. PMID 12121919
- [Background] Abruzzo GK, Flattery AM, Gill CJ, Kong L, Smith JG, Pikounis VB, Balkovec JM, Bouffard AF, Dropinski JF, Rosen H, Kropp H, Bartizal K. Evaluation of the echinocandin antifungal MK-0991 (L-743,872): efficacies in mouse models of disseminated aspergillosis, candidiasis, and cryptococcosis. Antimicrob Agents Chemother. 1997 Nov;41(11):2333-8. doi: 10.1128/AAC.41.11.2333. PMID 9371329
- [Background] Abruzzo GK, Gill CJ, Flattery AM, Kong L, Leighton C, Smith JG, Pikounis VB, Bartizal K, Rosen H. Efficacy of the echinocandin caspofungin against disseminated aspergillosis and candidiasis in cyclophosphamide-induced immunosuppressed mice. Antimicrob Agents Chemother. 2000 Sep;44(9):2310-8. doi: 10.1128/AAC.44.9.2310-2318.2000. PMID 10952573
- [Background] Bernard EM, Ishimaru T, Armstrong D. Low doses of the pneumocandin L-743,872, are effective for prevention and treatment in an animal model of pulmonary aspergillosis (abstract: 106). 36th Interscience Conference on Antimicrobial Agents and Chemotherapy; New Orleans, Louisiana, 1996.
- [Background] Graybill JR, Bocanegra R, Luther M, Fothergill A, Rinaldi MJ. Treatment of murine Candida krusei or Candida glabrata infection with L-743,872. Antimicrob Agents Chemother. 1997 Sep;41(9):1937-9. doi: 10.1128/AAC.41.9.1937. PMID 9303388
- [Background] Graybill JR, Najvar LK, Montalbo EM, Barchiesi FJ, Luther MF, Rinaldi MG. Treatment of histoplasmosis with MK-991 (L-743,872). Antimicrob Agents Chemother. 1998 Jan;42(1):151-3. doi: 10.1128/AAC.42.1.151. PMID 9449276
- [Background] Kohler S, Wheat LJ, Connolly P, Schnizlein-Bick C, Durkin M, Smedema M, Goldberg J, Brizendine E. Comparison of the echinocandin caspofungin with amphotericin B for treatment of histoplasmosis following pulmonary challenge in a murine model. Antimicrob Agents Chemother. 2000 Jul;44(7):1850-4. doi: 10.1128/AAC.44.7.1850-1854.2000. PMID 10858342
- [Background] Powles MA, Liberator P, Anderson J, Karkhanis Y, Dropinski JF, Bouffard FA, Balkovec JM, Fujioka H, Aikawa M, McFadden D, Schmatz D. Efficacy of MK-991 (L-743,872), a semisynthetic pneumocandin, in murine models of Pneumocystis carinii. Antimicrob Agents Chemother. 1998 Aug;42(8):1985-9. doi: 10.1128/AAC.42.8.1985. PMID 9687394
- [Background] Onishi J, Meinz M, Thompson J, Curotto J, Dreikorn S, Rosenbach M, Douglas C, Abruzzo G, Flattery A, Kong L, Cabello A, Vicente F, Pelaez F, Diez MT, Martin I, Bills G, Giacobbe R, Dombrowski A, Schwartz R, Morris S, Harris G, Tsipouras A, Wilson K, Kurtz MB. Discovery of novel antifungal (1,3)-beta-D-glucan synthase inhibitors. Antimicrob Agents Chemother. 2000 Feb;44(2):368-77. doi: 10.1128/AAC.44.2.368-377.2000. PMID 10639364
- [Background] Hajdu R, Thompson R, Sundelof JG, Pelak BA, Bouffard FA, Dropinski JF, Kropp H. Preliminary animal pharmacokinetics of the parenteral antifungal agent MK-0991 (L-743,872). Antimicrob Agents Chemother. 1997 Nov;41(11):2339-44. doi: 10.1128/AAC.41.11.2339. PMID 9371330
- [Background] Stone JA, Holland SD, Wickersham PJ, Sterrett A, Schwartz M, Bonfiglio C, Hesney M, Winchell GA, Deutsch PJ, Greenberg H, Hunt TL, Waldman SA. Single- and multiple-dose pharmacokinetics of caspofungin in healthy men. Antimicrob Agents Chemother. 2002 Mar;46(3):739-45. doi: 10.1128/AAC.46.3.739-745.2002. PMID 11850256
- [Background] Stone EA, Fung HB, Kirschenbaum HL. Caspofungin: an echinocandin antifungal agent. Clin Ther. 2002 Mar;24(3):351-77; discussion 329. doi: 10.1016/s0149-2918(02)85039-1. PMID 11952021
- [Background] Balani SK, Xu X, Arison BH, Silva MV, Gries A, DeLuna FA, Cui D, Kari PH, Ly T, Hop CE, Singh R, Wallace MA, Dean DC, Lin JH, Pearson PG, Baillie TA. Metabolites of caspofungin acetate, a potent antifungal agent, in human plasma and urine. Drug Metab Dispos. 2000 Nov;28(11):1274-8. PMID 11038152
- [Background] . Stone JA, Holland S, Li S, et al. Effect of hepatic insufficiency on the pharmacokinetics of caspofungin (abstract: 14). 41st Interscience Conference on Antimicrobial Agents and Chemotherapy, Chicago, Illinois, 2001
- [Background] Stone JA, Holland S, Wickersham P, et al. Drug interaction between caspofungin and tacrolimus (abstract: 13). 41st Interscience Conference on Antimicrobial Agents and Chemotherapy, Chicago, Illinois, 2001.
- [Background] Villanueva A, Arathoon EG, Gotuzzo E, Berman RS, DiNubile MJ, Sable CA. A randomized double-blind study of caspofungin versus amphotericin for the treatment of candidal esophagitis. Clin Infect Dis. 2001 Nov 1;33(9):1529-35. doi: 10.1086/323401. Epub 2001 Oct 4. PMID 11588698
- [Background] Arathoon EG, Gotuzzo E, Noriega LM, Berman RS, DiNubile MJ, Sable CA. Randomized, double-blind, multicenter study of caspofungin versus amphotericin B for treatment of oropharyngeal and esophageal candidiases. Antimicrob Agents Chemother. 2002 Feb;46(2):451-7. doi: 10.1128/AAC.46.2.451-457.2002. PMID 11796357
- [Background] Villanueva A, Gotuzzo E, Arathoon EG, Noriega LM, Kartsonis NA, Lupinacci RJ, Smietana JM, DiNubile MJ, Sable CA. A randomized double-blind study of caspofungin versus fluconazole for the treatment of esophageal candidiasis. Am J Med. 2002 Sep;113(4):294-9. doi: 10.1016/s0002-9343(02)01191-9. PMID 12361815
- [Background] Mora-Duarte J, Betts R, Rotstein C, Colombo AL, Thompson-Moya L, Smietana J, Lupinacci R, Sable C, Kartsonis N, Perfect J; Caspofungin Invasive Candidiasis Study Group. Comparison of caspofungin and amphotericin B for invasive candidiasis. N Engl J Med. 2002 Dec 19;347(25):2020-9. doi: 10.1056/NEJMoa021585. PMID 12490683
- [Background] Maertens J, Raad I, Sable CA, et al. Multicenter, noncomparative study to evaluate safety and efficacy of caspofungin in adults with invasive aspergillosis refractory or intolerant to amphotericin B, amphotericin B lipid formulations, or azoles (abstract). 40th Interscience Conference on Antimicrobial Agents and Chemotherapy; Toronto, Canada, 2000
- [Background] Hiemenz JW, Raad II, Maertens JA, Hachem RY, Saah AJ, Sable CA, Chodakewitz JA, Severino ME, Saddier P, Berman RS, Ryan DM, Dinubile MJ, Patterson TF, Denning DW, Walsh TJ. Efficacy of caspofungin as salvage therapy for invasive aspergillosis compared to standard therapy in a historical cohort. Eur J Clin Microbiol Infect Dis. 2010 Nov;29(11):1387-94. doi: 10.1007/s10096-010-1013-0. Epub 2010 Aug 12. PMID 20703506
- [Background] . Maertens J, Raad I, Petrikkos G, et al. Update of the multicenter, noncomparative study of caspofungin in adults with invasive aspergillosis refractory or intolerant to other antifungal agents: an analysis of 90 patients (abstract). 42th Interscience Conference on Antimicrobial Agents and Chemotherapy; San Diego, California, USA, 2002.
- [Background] Ascioglu S, Rex JH, de Pauw B, Bennett JE, Bille J, Crokaert F, Denning DW, Donnelly JP, Edwards JE, Erjavec Z, Fiere D, Lortholary O, Maertens J, Meis JF, Patterson TF, Ritter J, Selleslag D, Shah PM, Stevens DA, Walsh TJ; Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Mycoses Study Group of the National Institute of Allergy and Infectious Diseases. Defining opportunistic invasive fungal infections in immunocompromised patients with cancer and hematopoietic stem cell transplants: an international consensus. Clin Infect Dis. 2002 Jan 1;34(1):7-14. doi: 10.1086/323335. Epub 2001 Nov 26. PMID 11731939
- [Background] Rex JH, Walsh TJ, Sobel JD, Filler SG, Pappas PG, Dismukes WE, Edwards JE. Reply to Dr. Chandrasekar (Clin Infect Dis 2001; 32:320-1) and Drs. Marr and Boeckh (Clin Infect Dis 2001; 32:321). Clin Infect Dis. 2001 Feb 1;32(3):518-9. doi: 10.1086/318517. No abstract available. PMID 11170965
- [Background] Stevens DA, Kan VL, Judson MA, Morrison VA, Dummer S, Denning DW, Bennett JE, Walsh TJ, Patterson TF, Pankey GA. Practice guidelines for diseases caused by Aspergillus. Infectious Diseases Society of America. Clin Infect Dis. 2000 Apr;30(4):696-709. doi: 10.1086/313756. Epub 2000 Apr 20. PMID 10770732
- See also: Related Info — http://www.aehh.org